CLINICAL TRIAL: NCT06202053
Title: Modified Uniportal Periareolar Incision Versus Conventional Uniportal Video-assisted Thoracic Surgery for Pulmonary Nodules: Protocol for a Prospective, Randomized, Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Union-99
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-01

CONDITIONS: Surgical Incision; Minimally Invasive Surgery
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (patients who received modified periareolar incision) (Experimental)
  Interventions: Procedure: Type of surgical incision
- Control group (patients who received conventional uniportal thoracoscopic incision) (No Intervention)

INTERVENTIONS:
Procedure: Type of surgical incision — The experimental group (patients received periareolar incision):
  An arc-shaped incision was made on the lateral side of the patient's affected areola. The subcutaneous tissue was then dissociated between the lateral mammary gland and the skin to the level of the fourth intercostal space in front of the midaxillary line. The fatty tissue behind the breast was separated horizontally to expose the serratus anterior muscle, and an intercostal incision was made. The skin was pulled back throughout the procedure to expose a better surgical field and avoid damage to the mammary gland.
  The control group (patients underwent an axillary incision):
  For patients in the control group, an incision was made into the fourth intercostal space in the midline of the axilla, where subcutaneous tissue was separated and entered the chest.
  Arms: Experimental group (patients who received modified periareolar incision)

SUMMARY:
Minimally invasive surgical techniques, including the uniportal approach, have become widely adopted in thoracic surgery. Both surgeons and patients aim to achieve incisions that are as minimally invasive and cosmetically favorable as possible. However, achieving the ideal uniportal incision remains challenging, as some patients inevitably experience complications such as scar hyperplasia or incision depression. Increasing expectations for superior surgical outcomes and improved postoperative quality of life place additional demands on thoracic surgeons. The periareolar approach, although rarely reported, typically involves entering the chest cavity directly through the mammary gland. Its application has been limited in the literature. In this study, we modified the periareolar incision by establishing a subcutaneous tunnel to minimize damage to the mammary gland. We aim to assess the feasibility and safety of this modified periareolar incision as a novel option for uniportal thoracoscopic surgery.Participants were divided into two groups: the modified periareolar incision group and the conventional uniportal video-assisted thoracic surgery (VATS) group. In the modified periareolar incision group, a curved incision was made along the lateral areola of the affected side. A subcutaneous tunnel was created between the mammary gland and the skin, extending to the fourth or fifth intercostal space along the anterior midaxillary line, where an intercostal incision was performed to access the thoracic cavity. In the conventional uniportal VATS group, patients were directly accessed through an intercostal incision in the midaxillary line. The primary endpoints of the study were the incidence of postoperative complications and the rate of conversion to thoracotomy during the operation. Postoperative complications were monitored and recorded for up to 3 months after surgery. The secondary endpoints of the study were differences in postoperative pain scores and cosmetic satisfaction between the two groups. Additional analyses included baseline patient characteristics and operative data. Postoperative pain was assessed using the Visual Analogue Scale (VAS) on postoperative days 1, 2, 3, and 7. Incision recovery was evaluated at 1 and 3 months post-surgery using the Patient and Observer Scar Assessment Scale (POSAS). Cosmetic satisfaction with the incision was assessed 1 month postoperatively using a 5-point scale (1 = very dissatisfied; 5 = very satisfied). Patients were also presented with photos of two incision types and asked to choose their preferred style. Modified periareolar incision is a small improvement of previously reported incision, but it significantly increases the number of procedures available and the number of patients who can be included. The modified periareolar incision could be used as a new option for uniportal VATS segmentectomy, and it was more cosmetic and less invasive,

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients aged 18-75 years
2. Good degree of movement of the areola (being able to move to the anterior axillary line)
3. Meeting the criteria for thoracoscopic surgery, including lobectomy (expected absence of adhesions, well-developed interlobar fissure) and sublobectomy (including segmentectomy and wedge resection)
4. No evidence of advanced lung cancer on preoperative evaluation
5. No history of chemotherapy, immunotherapy, or radiotherapy
6. ECOG performance status 0-1;
7. Patients and their families agreed to participate in this study and signed a written informed consent form.

Exclusion criteria:

1. Patients had previously undergone pneumonectomy or preoperative chemotherapy and/or radiotherapy
2. Previous breast surgery
3. Risk of conversion to thoracotomy or changing the incision during the operation
4. Poor preoperative lung function
5. Presence of other cancers or other advanced diseases
6. Preoperative pulmonary infection or uncontrolled acute pulmonary disease or acute exacerbation of chronic obstructive pulmonary disease
7. Severe hypertension (resting systolic/diastolic blood pressure of >180/100 mmHg), intracranial mass, or intracranial hypertension
8. Recent brain injury, cerebral infarction, or cerebral hemorrhage
9. Hyperthyroidism
10. Previous history of angina pectoris, myocardial infarction, or heart failure
11. History of thoracoscopic resection of mediastinal and pleura tumors
12. Central nervous system disease; mental or neurological diseases, cognitive or language dysfunction due to which the patient was unable to cooperate with the follow-up
13. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 1 month after the operation
  Patients were followed up after surgery for complications
Rate of conversion to thoracotomy during the operation. | During surgery

SECONDARY OUTCOMES:
Postoperative pain score | 1 week after the operation
  Postoperative pain was assessed using the Visual Analogue Scale (VAS) on postoperative days 1, 2, 3, and 7
Cosmetic satisfaction with the incision | 1 month after the operation
  Cosmetic satisfaction with the incision was assessed 1 month postoperatively using a 5-point scale (1 = very dissatisfied; 5 = very satisfied). Patients were also presented with photos of two incision types and asked to choose their preferred style
Incision recovery | 3 months post-surgery
  Incision recovery was evaluated at 1 and 3 months post-surgery using the Patient and Observer Scar Assessment Scale (POSAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China